CLINICAL TRIAL: NCT00794209
Title: Phase lb, Five Period Crossover, Open-Label Study Evaluating a Single Dose Administration of 3mL or 5mL of Inhaled AeroLEF (Liposome-Encapsulated Fentanyl 500 Mcg/mL), Delivered by up to Four Aerosol Delivery Devices in Healthy Subjects
Brief Title: Study Evaluating Inhaled AeroLEF Delivered in 4 Aerosol Delivery Devices in Healthy Volunteers
Acronym: LEF-07
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Responsible Party: Ali Raza, YM BioSciences
Model: Crossover | Masking: None
Other Study IDs: LEF-07
Record Dates: First submitted 2008-11-13; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: AeroLEF, fentanyl, liposome encapsulated, opioid
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: i.v fentanyl, AeroLEF

INTERVENTIONS:
Drug: i.v fentanyl, AeroLEF — * i.v fentanyl
  * 5 mL of AeroLEF in Opti-Mist 750E continuous flow nebulizers (Maersk Medical Inc., (USA), McAllen, Texas)
  * 5 mL, of AeroLEF in Misty-Neb continuous flow nebulizers (Allegiance Healthcare Corp., McGaw Park, Illinois)
  * 5 mL of AeroLEF in PARI LC-Plus continuous flow nebulizers (PARI Respiratory Equipment Inc., London, Ontario)
  * 3 mL, of AeroLEF in AeroEclipse breath-actuated nebulizers (Trudell Medical International, London, Ontario) - reference device.
  Other Names: fentanyl, AeroLEF

SUMMARY:
This was an open-label, two-phase, crossover, safety, pharmacokinetic (PK), and pharmacodynamic (PD) study in normal, healthy, non-smoking, fasting male and female subjects. The first phase (A. Device Qualification Phase) of the study compared three aerosol devices to a reference device to identify a nebulizer that produced a favourable, clinically relevant, PK and PD profile of AeroLEF. The PK and PD of the test and reference devices were compared to 200 mcg of intravenous fentanyl administered over 1 minute.

The second phase (B. Device Characterization Phase) of the study was planned to characterize and compare the safety, PK and PD of the selected aerosol device (identified in the Device Qualification Phase) to 300mcg of intravenous fentanyl administered over 15 minutes if a device was chosen during the Device Qualification Phase. The data from the selected aerosol device would be pooled from subjects in both the Device Qualification and Device Characterization Phases of the study.

DETAILED DESCRIPTION:
A. Device Qualification Phase The Device Qualification Phase was an open-label, five-period, crossover design. Subjects received one dose (5mL) of inhaled AeroLEF (500 mcg/mL as fentanyl base) as administered by the Opti-Mist continuous flow jet nebulizer (test device), one dose (5mL) of inhaled AeroLEF (500 mcg/mL as fentanyl base) as administered by the Misty-Neb continuous flow jet nebulizer (test device), one dose (5mL) of inhaled AeroLEF (500 mcg/mL as fentanyl base) as administered by the PARI-LC Plus continuous flow jet nebulizer (test device), and one dose (3mL) of inhaled AeroLEF (500 mcg/mL as fentanyl base) as administered by the AeroEclipse breath-actuated nebulizer (reference device) in treatment sessions 1, 2, 3, and 5. A washout period of at least 7 days separated each of the dosing sessions.

In the fourth treatment session (session 4), subjects received a single dose of intravenous Fentanyl Citrate USP (200 mcg) administered over 1 minute, following a washout period of at least 7 days after the previous study treatment. This session was conducted while the data analysis for device qualification was proceeding, as the results from the fourth session were not required for the data analysis.

Nine (9) subjects participated in the following study visits in order to maintain group sizes of 6 volunteers per session: pre-study screening (two visits within 28 days prior to the first dose), treatment period (five visits) and follow-up (one visit 7-14 days following last dosing session). Each visit involving pharmacokinetic, pharmacodynamic and safety assessments was scheduled for each individual at approximately the same time of day.

The pre-study screening visits confirmed the eligibility for the study, and trained subjects in the use of nebulizer devices and the pupillometry procedures. Subjects continued in the study if they were comfortable using the nebulizer devices, and the pupillometry measurement system could reliably measure their pupils.

For each of the treatment sessions, study drug was administered on the morning of the treatment day, and blood collections and pupillometry assessments were performed to generate a pharmacokinetic and pharmacodynamic profile from immediately prior to dosing to approximately 24 hours following dosing. Adverse events were documented throughout the treatment sessions. A safety assessment was performed prior to discharge from the clinic at about 24 hours post-dose.

B. Device Characterization Phase This was planned to be an open-label, two-period, crossover, safety, pharmacokinetic, and pharmacodynamic design in normal, healthy, non-smoking, fasting male and female subjects. Subjects who participated in the Device Qualification Phase were to not eligible to participate in the Device Characterization Phase.

Subjects would have received one dose (5 mL) of inhaled AeroLEF (500 mcg/mL of fentanyl base) as administered by the continuous flow nebulizer device, Opti-Mist, Misty-Neb or PARI LC-Plus, selected in the Device Qualification Phase of the study. In a second treatment session, subjects would have received a single dose of 300 mcg of intravenous Fentanyl Citrate USP administered over 15 minutes. A washout period of at least 7 days was planned to separate the two dosing sessions.

Subjects would have participated in similar study visits as described for the Device Qualification Phase: pre-study screening (two visits within 28 days prior to the first dose), treatment phase (two visits), and follow-up (one visit). Pharmacokinetic, pharmacodynamic, and safety parameters would have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 65 years, inclusive. No history of smoking for greater than or equal to 12 months, and no smoking within the past year by self-report.
2. Body weight with a Body Mass Index (BMI) range of 18.5 -- 27.0, with a minimum weight of at least 60 kg.
3. Normal findings in the physical examination and vital signs (blood pressure between 100-150/60-90 mmHg, heart rate between 55-99 beats, respiration 12--24/min) and no clinically significant findings in a 12-lead electrocardiogram (ECG).
4. Negative urine screen for drugs of abuse.
5. Negative tests for smoking tobacco (carbon monoxide (CO) breath test), alcohol (breath test), hepatitis B-surface antigen, hepatitis C antibody, and HIV at screening.
6. No clinical laboratory values outside of the laboratory normal reference range, unless the Principal Investigator decided they were not clinically significant.
7. Female subjects: (a) if pre-menopausal, and were not pregnant prior to study start and would avoid pregnancy during the study and up until one (1) month after the end of the study by the use of adequate contraceptive precautions (abstinence or the use of two effective methods, e.g. oral contraceptive pill and condom with spermicidal foam), or (c) were surgically sterile for at least 6 months, or (d) post-menopausal for at least 1 year.
8. Female subjects of childbearing potential must have negative pregnancy tests at screening (serum test) and prior to dosing at each treatment session (urine test).
9. Ability and willingness to communicate well with the investigator and to comply with the requirements of the entire study.
10. Willingness to give written informed consent (prior to any study-related procedures being performed) and was able to adhere to the study restrictions, appointments, and examination schedule.

Exclusion Criteria:

1. Known history of hypersensitivity to fentanyl (e.g. Fentanyl citrate, Actiq, Duragesic, Sublimaze®) and/or related opioid analgesic drugs such as: alfentanil HC1 (Rapifen®), amleridine, butorphanol tartrate (Stadol NSA®), codeine (Tylenol® No. 3), hydrocodone (Tussionex®, Hycodan®, Hycomine®), hydromorphone (Dilaudid®), methadone, morphine (MS Contin®), nalbuphine (Nubain®}, oxycodone (Percocet®, Percodan®, oxymorphone (Numorphan®), pentazocine (Talwin®), pethidine, meperidine (Demerol®), propoxyphene (Darvon®, dextropropoxyphene), remifentanil (Ultiva®), or sufentanil.
2. History of violent behaviour under the influence of opioids.
3. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, neuromuscular, neurological, hematological, liver or kidney disease, or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
4. Known history of chronic bronchitis or other bronchospastic condition.
5. Any known nasal cavity abnormality or aversion to this route of drug administration.
6. History of glaucoma or any other pupil abnormalities that, in the opinion of the Principal Investigator, would interfere with the ability to perform the pupillometry measurements.
7. Any clinically significant illness during the last four (4) weeks prior to entry into this study which, in the opinion of the Principal Investigator, would introduce additional risk for the study subject, or was likely to interfere with the successful collection of the measures required.
8. Presence of any significant physical or organ abnormality that, in the opinion of the Principal Investigator, would introduce additional risk for the study subject, or was likely to interfere with the successful collection of the measures required.
9. Any subject with a lifetime history of dependency on opiates by DSM-IVr criteria or any other drugs of abuse.
10. Any current major is I psychiatric disorder for which the subject was currently receiving treatment or which would make study compliance an issue, or a history of severe neurological disease, such as head injury or recurrent seizures.
11. Use of any prescription medication within 30 days preceding entry into this study, including any enzyme-inducing or enzyme-inhibiting drugs (with the exception of oral, depot or injectable contraceptives for women).
12. Use of over-the-counter (OTC) medication within 14 days preceding entry into this study (excluding OTC products known to not affect the cytochrome P450 system, and OTC contraceptive products).
13. Participation in a clinical trial with an investigational drug within 30 days preceding this study.
14. Subjects who received treatment in the Device Qualification Phase of this study was to be excluded from participation in the Device Characterization Phase of this study.
15. Blood donation or other blood draws within 45 days prior to enrolment in the study resulting in a total withdrawal of 100 mL or greater.
16. Significant or recent history of asthma (after 12 years of age).
17. Any subject with a recent (less than 1 year) history of alcohol dependency.
18. History of hiatus hernia, reflux disease or gastroesophageal reflux disease (GERD).
19. Inability to tolerate abstinence from caffeine for 48 hours prior to and during each of the study treatment phases.
20. Any condition, for which the study or participation in the study would pose a safety risk to the subject.
21. History of serious adverse reaction or hypersensitivity to any drug.
22. Females who were lactating or at risk of pregnancy (i.e., sexually active and not using an adequate form of birth control).
23. Inability to reliably generate a pupil measurement, inability to perform reproducible spirometry (based on FEV1), inability to adequately or comfortably use the nebulizer devices on the Study Procedures Training and Qualification Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-03; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
To identify an aerosol device which maintains the plasma fentanyl concentration above the lower limit of the therapeutic range (> 0.5 ng/mL) for at least 2 hours longer than the AeroEclipse breath-actuated nebulizer | duration of 2 months

SECONDARY OUTCOMES:
To characterize and compare the pharmacokinetic, pharmacodynamic and safety profiles of single inhaled doses of AeroLEF (liposome encapsulated fentanyl, 500 mcg/mL) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Sellers, MD, Principal Investigator — Ventana Clinical Research Corporation